CLINICAL TRIAL: NCT05596253
Title: Incidence and Predictors of Post-TIPS (Transjugular Intrahepatic Portosystemic Shunt (TIPS) Heart Failure in Patients With Cirrhosis
Brief Title: Incidence and Predictors of Post-TIPS Heart Failure in Patients With Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, MD, West China Hospital
Other Study IDs: HF-TIPS
Record Dates: First submitted 2022-10-23; First posted 2022-10-27 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Liver Cirrhosis; Transjugular Intrahepatic Portosystemic Shunt (TIPS); Heart Failure
MeSH Terms: conditions — Liver Cirrhosis; Heart Failure | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cirrhosis who underwent TIPS: Patients with cirrhosis who underwent TIPS due to complications of portal hypertension were inclueded for observation.
  Interventions: Procedure: TIPS

INTERVENTIONS:
Procedure: TIPS — TIPS: Established distributary channel between the portal vein and hepatic vein via the jugular vein, portal vein blood directly shunts into the systemic circulation to reduce portal vein pressure to effectively prevent bleeding and refractory ascites.

SUMMARY:
The purpose of this study is to conduct a prospective trial to investigate the incidence of heart failure in cirrhosis patients undergoing transjugular intrahepatic portosystemic shunt ,and to analyze the the predictors and modififications of cardiac function.

DETAILED DESCRIPTION:
Hyperdynamic circulation is a common Phenomenon in cirrhosis due to systemic and splanchnic vasodilatation, which may result cardic dysfunction and abnormal structure ,called cirrhotic cardiomyopathy(CCM). Transjugular intrahepatic portosystemic shunt (TIPS), as a effective technique to alleviates portal hypertension in cirrhotic patients, often be used to treat with refractory ascites and variceal bleeding which endoscopy and drug therapy are ineffective. However, owing to the increased shunting of blood from the splanchnic vascular bed into the central vascular bed, TIPS further exacerbates the hyperdynamic circulatory state, which may lead to heart failure.yet there are no convincing research to study the incidence of heart failure in cirrhosis after transjugular intrahepatic portosystemic shunt. The purpose of this study is to conduct a prospective trial to investigate the incidence of heart failure in cirrhotic patients undergoing transjugular intrahepatic portosystemic shunt ,and to analyze the the predictors and modififications of cardiac function.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis
2. TIPS is placed successfully
3. Agree to participate in the trial

Exclusion Criteria:

1. Non-cirrhotic portal hypertension
2. Previous TIPS or surgical shunt
3. Medium to severe pulmonary hypertension
4. Heart failure
5. End-stage renal disease requiring hemodialysis
6. Respiratory failure
7. Malignancies with a life expectancy of less than 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cirrhotic patients undergoing TIPS
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of heart failue | up to 36 months
  Heart failue assessed by2021 ESC Guidelines

SECONDARY OUTCOMES:
Predictors of heart Failure | up to 36 months
  Heart failue assessed by2021 ESC Guidelines
mortality | up to 36 months
  Telephone follow-up was performed to collect relevant information
Modififications of cardiac function | up to 36 months
  Echocardiography was to evaluate cardic function

CONTACTS AND LOCATIONS:
Overall Officials: xuefeng luo, Principal Investigator — Sichuan University
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided